CLINICAL TRIAL: NCT02370407
Title: Assessment of the Transferability of Skills From Robotic to Laparoscopic Simulation Platforms in Surgical Skill Naive Participants
Brief Title: Assessment of the Transferability of Skills From Robotic to Laparoscopic Simulation Platforms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00031436
Record Dates: First submitted 2014-11-25; First posted 2015-02-24 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Surgical Simulation Education
Keywords: surgical education; minimally invasive surgical procedures; laparoscopic simulation; robotic simulation; medical education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic simulator (Experimental): 20 study participants will be randomized to perform peg transfer task on a laparoscopic simulator 10 times (Fundamentals of Laparoscopic Surgery (FLS), VT Medical Inc, Waltham, MA).
  Interventions: Device: a laparoscopic simulator (Fundamentals of Laparoscopic Surgery (FLS), VT Medical Inc, Waltham, MA)
- Mimic da Vinci robotic simulator (Experimental): 20 study participants will be randomized to perform peg board 1 exercise 10 times on a Mimic da Vinci robotic simulator (Mimic da Vinci Simulator, Intuitive Surgical, Sunnyvale, CA).
  Interventions: Device: Mimic da Vinci robotic simulator

INTERVENTIONS:
Device: a laparoscopic simulator (Fundamentals of Laparoscopic Surgery (FLS), VT Medical Inc, Waltham, MA) — 10 repetitions of practice on laparoscopic simulator.
  Arms: Laparoscopic simulator
Device: Mimic da Vinci robotic simulator — 10 repetitions of practice on Mimic da Vinci robotic simulator.
  Arms: Mimic da Vinci robotic simulator

SUMMARY:
This is a randomized controlled trial that will randomize 40 surgical skill naive medical students to practice on a robotic simulator or laparoscopic simulator after first completing a baseline evaluation on both surgical simulation platforms. Medical students will be evaluated again after 10 practice sessions on the laparoscopic or robotic platforms to assess transferability of skills between the surgical simulation platforms.

DETAILED DESCRIPTION:
This is a randomized controlled trial that will randomize medical students to practice on a robotic simulator or a laparoscopic simulator. The investigators will first obtain baseline data by having the study participants perform one task (peg transfer exercise) on a laparoscopic simulator (Fundamentals of Laparoscopic Surgery (FLS), VT Medical Inc, Waltham, MA), and a similar task on a robotic trainer (Mimic da Vinci Simulator, Intuitive Surgical, Sunnyvale, CA). Participants will then be randomized to practice on the robotic simulator or practice on the laparoscopic trainer for at least 10 repetitions. After the participants complete 10 repetitions, they will be evaluated again on both the laparoscopic and robotic simulator using time to task completion and Mimi DV trainer motion metrics. Two expert laparoscopic and robotic surgeons will also evaluate participant performance using previously validated global rating scales for robotic and laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Medical students with no prior laparoscopic or robotic experience in clinical or practice setting

Exclusion Criteria:

* Prior laparoscopic or robotic experience in clinical setting or in practice setting

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi Chiung Grace Chen, MD, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Derived] Orlando MS, Thomaier L, Abernethy MG, Chen CCG. Retention of laparoscopic and robotic skills among medical students: a randomized controlled trial. Surg Endosc. 2017 Aug;31(8):3306-3312. doi: 10.1007/s00464-016-5363-2. Epub 2017 Jan 11. PMID 28078455

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laparoscopic Simulator | Mimic da Vinci Robotic Simulator
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Simulator | Mimic da Vinci Robotic Simulator | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Time to Task Completion (Robotic Task)
Description: Primary outcome will be time to task completion (seconds) on the robotic task
Time Frame: 1 day of practice
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Laparoscopic Group: Training on laparoscopic platform resulted in improved performance on laparoscopic and robotic task
- Robotic Group: Training on robotic platform resulted in improved performance on laparoscopic and robotic task
Arm/Group | Laparoscopic Group | Robotic Group
Number analyzed (Participants) | 20 | 20
seconds | 120 (42) | 71 (23)

2. Primary Outcome: Global Rating Scale Score on the Laparoscopic Task
Description: Global rating scale score on the laparoscopic task. A composite score of (1) depth perception, (2) bimanual dexterity, (3) efficiency, (4) tissue handling, (5) time and motion, (6) instrument handling, and (7) flow of operation, each scored 1 through 5 on an anchored Likert scale where higher scores indicated improved proficiency. Point range 7 - 35.
Time Frame: Study duration
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Laparoscopic: 10 repetitions on laparoscopic task
- Robotic: 10 repetitions on robotic task
Arm/Group | Laparoscopic | Robotic
Number analyzed (Participants) | 20 | 20
units on a scale | 22.5 (3.8) | 16.3 (4.1)

3. Primary Outcome: Global Rating Scale Score on the Robotic Task
Description: A composite score of (1) depth perception, (2) bimanual dexterity, (3) efficiency, (4) tissue handling, (5) time and motion, (6) instrument handling, and (7) flow of operation, each scored 1 through 5 on an anchored Likert scale where higher scores indicated improved proficiency. Point range 7 - 35.
Time Frame: Study duration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laparoscopic | Robotic
Number analyzed (Participants) | 20 | 20
units on a scale | 16.9 (5.4) | 23.5 (6.7)

4. Primary Outcome: Time to Task Completion on the Laparoscopic Task
Description: Time to task completion (seconds) on the laparoscopic task
Time Frame: 1 day of practice
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Laparoscopic Group | Robotic Group
Number analyzed (Participants) | 20 | 20
seconds | 100 (29) | 158 (65)

5. Secondary Outcome: Economy of Motion on the Robotic Task
Description: (cm, where lower measurements represent improved economy of motion). This measures how many cm the instruments traveled in order to accomplish the task
Time Frame: Study duration
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Laparoscopic: 10 repetitions on the laparoscopic task
- Robotic Task: 10 repetitions on the robotic task
Arm/Group | Laparoscopic | Robotic Task
Number analyzed (Participants) | 20 | 20
cm | 241 (57) | 161 (35)

6. Secondary Outcome: Instrument Out of View
Description: Automatically recorded data on the Mimic DV trainer, (sec). The longer out of view indicates decreased proficiency
Time Frame: through study completion
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Laparoscopic Group | Robotic Group
Number analyzed (Participants) | 20 | 20
seconds | 3.06 (3.3) | 0.91 (2.3)

7. Secondary Outcome: Instrument Collisions
Description: Automatically recorded data on the Mimic DV trainer which records number of collisions
Time Frame: study duration
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Laparoscopic Group | Robotic Group
Number analyzed (Participants) | 20 | 20
number of events | 2.8 (4.3) | 1.1 (1.8)

8. Secondary Outcome: Time Spent Using Excessive Force
Description: Automatically recorded data on the Mimic DV trainer (seconds)
Time Frame: study duration
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Laparoscopic Group | Robotic Group
Number analyzed (Participants) | 20 | 20
seconds | 0.28 (0.58) | 0.24 (1.1)

9. Secondary Outcome: Workspace Range
Description: Automatically recorded data on the Mimic DV trainer consisting of workspace range (cm, this is the widest range traveled by the 2 instruments, one in each hand), and number of peg drops
Time Frame: study duration
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Laparoscopic Group | Robotic Group
Number analyzed (Participants) | 20 | 20
cm | 9.41 (2.3) | 9.34 (2.5)

ADVERSE EVENTS:
Description: 40 surgical skill naive medical students practiced techniques on simulators. They were randomized to either practice on a robotic simulator or laparoscopic simulator. No participants were at risk for health outcomes, as they were assessed only on time to completion of a task compared to the two different interventions. However, this was done only in a simulated setting, and not on a patient.
Groups:
- Laparoscopic Simulator: 20 study participants will be randomized to perform peg transfer task on a laparoscopic simulator 10 times (Fundamentals of Laparoscopic Surgery (FLS), VT Medical Inc, Waltham, MA).
  Laparoscopic simulator (Fundamentals of Laparoscopic Surgery (FLS), VT Medical Inc, Waltham, MA): 10 repetitions of practice on laparoscopic simulator.
Arm/Group | Laparoscopic Simulator | Mimic da Vinci Robotic Simulator
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
We modified three previously validated scales to create a 35-point scale to evaluate participants; therefore, the validity of these scales may have been impacted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No